CLINICAL TRIAL: NCT06544785
Title: A Multicenter, Phase 2 Randomized, Open Label Study to Evaluate Zanubrutinib in Combination With Obinutuzumab in Previously Untreated Patients With Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL) (GELLC-10-ZANUBIO)
Brief Title: Zanubrutinib With Obinutuzumab in Untreated Patients With Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GELLC-10-ZANUBIO
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: zanubrutinib; obinutuzumab; untreated CLL/SLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — zanubrutinib; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm Zanubrutinib+early Obinutuzumab (Experimental): Patients will be treated with the combination of zanubrutinib 320 mg P.O qDay and obinutuzumab, starting obinutuzumab at cycle 2 to reduce infusion-related reactions. Intravenous obinutuzumab will be given on days 1 (100 mg), 2 (900 mg), 8 (1000 mg), and 15 (1000 mg) of cycle 2 and on day 1 (1000 mg) of cycles 3-7.
  Response will be assessed after 20 cycles of treatment for the primary objective of the study. Patients that in the evaluation of cycle 20 who achieve uMRD will stop treatment with zanubrutinib, whereas the rest of patients will continue on treatment with zanubrutinib until progression, unacceptable toxicity or trial completion, whichever comes first. Patients who achieve an uMRD in bone marrow beyond C20, will also be allowed to stop the treatment, whereas the rest of patients will continue on treatment with zanubrutinib until progression, unacceptable toxicity, or trial completion, whichever comes first.
  Interventions: Drug: Zanubrutinib Oral Product; Drug: Obinutuzumab
- Arm Zanubutinib+late Obinutuzumab (Experimental): Patients will start treatment with zanubrutinib 320 mg P.O qDay in monotherapy. After 12 cycles of zanubrutinib patients will be treated with the combination of zanubrutinib and obitnutuzumab. Intravenous obinutuzumab will be given on days 1 (100 mg), 2 (900 mg), 8 (1000 mg), and 15 (1000 mg) of cycle 13 and on day 1 (1000 mg) of cycles 14-18.
  Response will be assessed after 20 cycles of treatment for the primary objective of the study. Patients that in the evaluation of cycle 20 who achieve uMRD will stop treatment with zanubrutinib, whereas the rest of patients will continue on treatment with zanubrutinib until progression, unacceptable toxicity or trial completion, whichever comes first. Patients who achieve an uMRD in bone marrow beyond C20, will also be allowed to stop the treatment, whereas the rest of patients will continue on treatment with zanubrutinib until progression, unacceptable toxicity, or trial completion, whichever comes first.
  Interventions: Drug: Zanubrutinib Oral Product; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Zanubrutinib Oral Product — Zanubrutinib drug product is supplied as 80 mg strengths in capsules for oral administration.
  In both arms A and B, zanubrutinib 320 mg will be taken qDay with or without food. Patients will take zanubrutinib with water at approximately the same time every day.
  Other Names: Zanubrutinib
Drug: Obinutuzumab — Each dose of obinutuzumab is 1000 mg administered intravenously, per institutional standards, with the exception of the first infusion in Cycle 2 (arm A) or Cycle 13 (arm B). It is recommended that the initial 1000 mg dose be administered over Day 1 (100 mg) and Day 2 (900 mg). For subjects who tolerate the initial 100 mg dose well and required no dose interruption or modification of the infusion rate, the treating physician may opt to administer the remaining 900 mg on Day 1.
  Arm A: patients will receive obinutuzumab on days 1 (100 mg), 2 (or day 1 continued, 900 mg), 8 and 15 (1000 mg) of the cycle 2 of zanubrutinib treatment, and on the day 1 of cycles 3-7 (1000 mg).
  Arm B: patients will receive obinutuzumab on days 1 (100 mg), 2 ( (or day 1 continued, 900 mg), 8 and 15 (1000 mg) of the cycle 13 of zanubrutinib treatment, and on the day 1 of cycles 14-18 (1000 mg).

SUMMARY:
The goal of this phase II randomized open label study is to compare the rate of complete remission (CR) with undetectable minimal residual disease (uMRD) obtained with zanubrutinib in combination with obinutuzumab with two different schedules of administration of obinutuzumab (starting obinutuzumab at cycle 2 or 12 months) in patients with previously untreated Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL). There is scarce information about which is the most appropriate schedule of combining the BTKi and the anti-CD20 monoclonal antibody, and whether treatment can be safely stopped in those patients attaining deep responses (CR with uMRD) remains to be determined.

Response will be assessed after 20 cycles of treatment for the primary objective of the study. Patients attaining uMRD will stop treatment with zanubrutinib, whereas the rest of patients will continue on treatment with zanubrutinib until progression, unacceptable toxicity, or trial completion, whichever comes first.

DETAILED DESCRIPTION:
This a multicenter, phase 2 randomized, open label study of the Spanish Group of CLL (GELLC) for patients with untreated CLL/SLL with 2 arms of treatment. In this study, 106 patients from 20 centers in Spain with untreated CLL/SLL will be randomized (1:1) to arm A (n= 53) or arm B (n= 53). The randomization will be stratified according to the presence/absence of deletion/mutation 17p/TP53 at the time of inclusion and based on the randomization list generated by the study statistician.

Arm A: Patients will be treated with the combination of zanubrutinib 320 mg P.O qDay and obinutuzumab, starting obinutuzumab at cycle 2 to reduce infusion-related reactions. Intravenous obinutuzumab will be given on days 1 (100 mg), 2 (900 mg), 8 (1000 mg), and 15 (1000 mg) of cycle 2 and on day 1 (1000 mg) of cycles 3-7.

Arm B: Patients will start treatment with zanubrutinib 320 mg P.O qDay in monotherapy. After 12 cycles of zanubrutinib patients will be treated with the combination of zanubrutinib and obitnutuzumab. Intravenous obinutuzumab will be given on days 1 (100 mg), 2 (900 mg), 8 (1000 mg), and 15 (1000 mg) of cycle 13 and on day 1 (1000 mg) of cycles 14-18.

Response will be assessed after 20 cycles of treatment for the primary objective of the study. Patients that in the evaluation of cycle 20 who achieve uMRD (<0.01% tumour cells by flow cytometry) will stop treatment with zanubrutinib, whereas the rest of patients will continue on treatment with zanubrutinib until progression, unacceptable toxicity or trial completion, whichever comes first. Patients who achieve an uMRD in bone marrow beyond C20, will also be allowed to stop the treatment, whereas the rest of patients will continue on treatment with zanubrutinib until progression, unacceptable toxicity, or trial completion, whichever comes first.

In addition, the efficacy and safety of the combination therapy with two different administration schedules of obinutuzumab will be analysed through the following outcome measures: i) Overall response rate, including Complete Remission (CR), CR with incomplete marrow recovery (CRi), Partial Remission (PR), and partial response with lymphocytosis; ii) MRD analysis; iiI) Duration of response and progression-free survival (PFS); iv) Safety: type, frequency, and severity of adverse events (AEs) and relationship of AEs to zanubrutinib or the combination of zanubrutinib and obinutuzumab; v) Response rate in relationship to molecular and genetic prognostic factors; vi) Immunological recovery; vii) Overall survival (OS); viii) Biomarkers for response.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with previously untreated CLL defined following IWCLL criteria (Hallek, 2018).
2. Must understand and voluntarily sign an informed consent form.
3. Age ≥ 18 years at the time of signing the informed consent form and must be able to adhere to the study visit schedule and other protocol requirements.
4. Must have a documented diagnosis of CLL or SLL [IWCLL guidelines for diagnosis and treatment of CLL (Hallek, 2018)] meeting at least one of the following criteria:

   * Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and/or thrombocytopenia.
   * Massive (i.e. ≥6 cm below the left costal margin) or progressive or symptomatic splenomegaly.
   * Massive nodes (i.e. ≥10 cm in longest diameter) or progressive or symptomatic lymphadenopathy.
   * Progressive lymphocytosis with an increase of ≥50% over a 2-month period, or lymphocyte doubling time (LDT) of less than 6 months.
   * A minimum of any one of the following disease-related symptoms: unintentional weight loss ≥ 10% within the previous 6 months, significant fatigue (i.e., ECOG PS 2 or worse; cannot work or unable to perform usual activities), fevers of greater than 38.0°C for 2 or more weeks without other evidence of infection, or night sweats for more than 1 month without evidence of infection.
   * Autoimmune complications including anemia or thrombocytopenia poorly responsive to corticosteroids.
   * Symptomatic or functional extranodal involvement (eg, skin, kidney, lung, spine).
5. Must have an Eastern Cooperative Oncology Group (ECOG) performance status score of ≤2.
6. Female patients of childbearing potential must practice highly effective methods of contraception initiated prior to first dose of study drug, for the duration of the study, and for ≥ 90 days after the last dose of zanubrutinib and 18 months after last dose of obinutuzumab.

   Male patients are eligible if vasectomized or if they agree to the use of barrier contraception with other applicable highly effective methods described below during the study treatment period and for ≥ 90 days after the last dose of zanubrutinib and 18 months after last dose of obinutuzumab.

   A woman is considered of childbearing potential, ie, fertile, following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. Contraception methods include the following:
   * Combined (estrogen- and progestogen- containing) hormonal contraception associated with the inhibition of ovulation - Oral, intravaginal, or transdermal.
   * Progestogen-only hormonal contraception associated with the inhibition of ovulation - Oral, injectable, implantable.
   * An intrauterine device.
   * Intrauterine hormone-releasing system.
   * Bilateral tubal occlusion.
   * Vasectomized partner (provided that the vasectomized partner is the sole sexual partner of the woman of childbearing potential study participant and that the vasectomized partner has received medical assessment of surgical success).
   * Sexual abstinence (defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment, starting the day prior to first dose of study drug, for the duration of the study, and for ≥ 90 days after the last dose of zanubrutinib or ibrutinib. Total sexual abstinence should only be used as a contraceptive method if it is in line with the patients' usual and preferred lifestyle. Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of exposure to investigational medicinal product, and withdrawal are not acceptable methods of contraception.

   Of note, barrier contraception (including male and female condoms with or without spermicide) is not considered a highly effective method of contraception, and, if used, this method must be used in combination with another acceptable method listed above.

   If patient is using hormonal contraceptives such as birth control pills or devices, a barrier method of contraception (eg, condoms) must also be used.

   A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle-stimulating hormone level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single follicle-stimulating hormone measurement is insufficient.
7. Female subjects of childbearing potential must have a negative pregnancy test at screening. Females of child bearing potential are defined as sexually mature women without prior hysterectomy or who have had any evidence of menses in the past 12 months. However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to other causes, including prior chemotherapy, anti-estrogens, or ovarian suppression.

Exclusion Criteria:

1. Prior treatment for CLL.
2. Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) and/or Hepatitis C Virus (HCV) infection. Subjects who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative could be eligible if they have an undetectable HBV DNA (negative polymerase chain reaction (PCR) <20 IU). Those who are hepatitis B surface antigen (HbsAg) positive or hepatitis B PCR positive will be excluded. Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded.

   Per published guidelines (NCCN 2012) or institutional guidelines, patients should be closely monitored for hepatitis B reactivation. Obtaining repeated hepatitis B PCR every 3 months during treatment and for the 12 months after last dose of study drug according to usual clinical practice in order to monitor for reactivation of hepatitis B is recommended.
3. Estimated Glomerular Filtration Rate (Cockcroft-Gault Appendix C) ≤30 mL/min/1.73m2.
4. Absolute neutrophil count (ANC) < 1.0 X 109/L.
5. Platelet count < 75 X 109/L, except for patients with bone marrow involvement by CLL in which case the platelet count must be ≥ 30 X 109/L.
6. Serum aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) or alanine transaminase (ALT)/serum glutamate pyruvate transaminase (SGPT) >2.5 x upper limit of normal (ULN).
7. Serum total bilirubin > 1.5 x ULN, except in cases of Gilbert's syndrome.
8. Prothrombin time/INR or aPTT (in the absence of Lupus anticoagulant) > 2x ULN.
9. Active bleeding, history of bleeding diathesis (eg, haemophilia or von Willebrand disease).
10. Unable to swallow capsules, or has disease significantly affecting gastrointestinal function that would limit absorption of oral medication.
11. Currently active, clinically significant cardiovascular disease or a history of myocardial infarction within 3 months prior to enrollment. Exception: Subjects with controlled, asymptomatic atrial fibrillation during screening can enrol on study.
12. Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon) within 7 days of first dose of study drug.
13. Systemic infection that has not resolved prior to initiating study treatment in spite of adequate anti-infective therapy.
14. Pregnant or lactating females.
15. Participation in any clinical study or having taken any investigational therapy within 28 days prior to initiating study therapy.
16. Central nervous system (CNS) involvement as documented by spinal fluid cytology or imaging.
17. Prior history of malignancies, other than CLL, unless the patient has been free of the disease for ≥ 3 years.

    Exceptions include the following:
    * Basal cell carcinoma of the skin
    * Squamous cell carcinoma of the skin
    * Carcinoma in situ of the cervix
    * Carcinoma in situ of the breast
    * Incidental histologic finding of prostate cancer (TNM stage of T1a or T1b)
18. Presence of autoimmune haemolytic anaemia or autoimmune thrombocytopenia.
19. Major surgery within the last 28 days prior to registration.
20. History of stroke or intracranial haemorrhage within 6 months prior to enrollment.
21. Requires treatment with strong CYP3A4/5 Inhibitors.
22. Known history of drug-specific hypersensitivity or anaphylaxis to study drug (including active product or excipient components).
23. Any life-threatening illness, medical condition, or organ system dysfunction which, in the Investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of zanubrutinib, or put the study outcomes at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2032-05-31 (Estimated); Study Completion 2032-05-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Complete Remission (CR) with undetectable Measurable Residual Disease (uMRD). | 7.5 Years
  To compare the rates of complete remission (CR) with undetectable minimal residual disease (uMRD, assessed by flow cytometry in bone marrow with a value <10-4 [0.01%] tumour cells for being considered as negative) between both arms A and B.
  Response will be assessed after 20 cycles of treatment for the primary outcome measure. Patients attaining uMRD will stop treatment with zanubrutinib, whereas the rest of patients will continue on treatment with zanubrutinib until progression, unacceptable toxicity, or trial completion, whichever comes first. Patients who achieve an uMRD in bone marrow beyond C20, will also be allowed to stop the treatment.
  The IWCLL guidelines (Hallek, 2018) will be used to measure response in CLL subjects.

SECONDARY OUTCOMES:
Overall response rate (ORR) | 7.5 Years
  Includes the following categories: Complete Remission (CR); CR with incomplete marrow recovery (CRi); Partial Remission (PR), and partial response with lymphocytosis.
  The IWCLL guidelines (Hallek, 2018) will be used to measure response in CLL subjects.
  Overall response assessment will include evaluation of physical exams, recording of symptoms, and haematological evaluations. OR will be assessed on Day 1 Cycle 2, on Day 1 of Cycles 3 to 12, and on Day 1 of Cycles 13, 15, 17, 19, 21, and 23, and then every 3 cycles to disease progression or study closure.
Measurable Residual Disease (MRD) analysis | 7.5 Years
  In cycle 20, MRD should be analysed in peripheral blood and in the bone marrow by flow-cytometry. Patients with uMRD should be followed every 6 months during 24 months and then every 12 months for MRD by peripheral blood flow cytometry. Patients with detectable MRD and without lymphocytosis (lymphocyte count < 4.0 X 109/L) should be followed every 6 months for MRD by peripheral blood flow cytometry during 24 months and then every 12 months. In addition, a further bone marrow MRD assessment should be performed at any time during follow-up when the patient has cleared MRD from the peripheral blood. MRD will also be evaluated in PB by flow-cytometry at cycle 9 in arm A (2 cycles after finalizing obinutuzumab).
Progression-Free Survival (PFS) | 7.5 Years
  Defined as the time from randomization until symptomatic disease progression (as defined by the updated iwCLL-guidelines) or death by any cause, whichever occurs first.
Overall Survival (OS) | 7.5 Years
  Defined as the time from the date of first dose of study drug to the date of the subject's death. If the subject is alive or the vital status is unknown, then the subject's data will be censored at the date the subject was last known to be alive.
  After progression, patients will be followed every 6 months to assess survival status and the start of subsequent cancer therapies until death, patient withdrawal, loss to follow-up, or study termination, whichever comes first.
Immunological recovery | 7.5 Years
  Serum quantitative immunoglobulin (IgG, IgM, IgA) levels will be evaluated by local laboratory at screening, on Day 1 of every odd cycle from Cycles 3 through 12, on Day 1 of every odd cycle (for Cycles 13, 15, 17, 19, 21 and 23), and then every 3 cycles until progression or study closure. The units if measure for the immunoglobulin levels determinations of will be g/L for all 3 Ig types.
Adverse Events (AE) | 7.5 Years
  Adverse Event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have a causal relationship with the treatment.
  Type, rate and severity of AEs and relationship of AEs to zanubrutinib or the combination of zanubrutinib and obinutuzumab, including the assessment of infusion related reactions (IRR) and tumour lysis syndrome (TLS) will be recorded. The rate and severity of IRR and TLS will be analyzed also according to the two different schedules of administration of obinutuzumab (arm A and arm B).

CONTACTS AND LOCATIONS:
Overall Officials: Pau Abrisqueta, Principal Investigator — Hospital Universitari Vall d'Hebrón; Francesc Bosch, Principal Investigator — Hospital Universitari Vall d'Hebrón
Locations (1):
- H. Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
All participant data relating to the study will be recorded on electronic CRF unless transmitted to the sponsor or designee electronically (e.g., laboratory data).
  The investigator is responsible for verifying that data entries are accurate and correct by physically or electronically signing the eCRF. Results of this clinical trial, positive or negative, will be presented at scientific conferences and published in scientific journals.